CLINICAL TRIAL: NCT04523701
Title: Diagnostic Role of the "White Test" With Lipidic Solution in the Early Intraoperative Identification of Open Bile Ducts for the Prevention of Bile Leakage After Liver Resection- A Randomized Controlled Multicentric Superiority Trial- The BiLe-Trial (Bile Leakage Trial)
Brief Title: Diagnostic Role of the "White Test" With Lipidic Solution in the Early Intraoperative Identification of Open Bile Ducts for the Prevention of Bile Leakage After Liver Resection (BiLe -Trial)
Acronym: BiLe
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Giulia Manzini (Other)
Responsible Party: Sponsor-Investigator, Giulia Manzini, Dr. med., Senior physician, Department of Visceral Surgery, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-02081; ex20Manzini
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Bile Leakage
Keywords: Liver resection; SMOFlipid 20%; White Test

STUDY DESIGN:
Intervention Model Description: Prospective randomized, controlled, observer and patient blinded multicentric (4 centres) superiority trial with 2 parallel study groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, care providers and outcome assessors are blinded, the surgical team is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (treatment) (Experimental): Open bile ducts are identified by visual control of the liver resection surface combined with the direct injection in the cystic stump of 20-40ml of SMOFlipid 20% Fresenius Kabi Canada Ltd.; authorization number: 57231 (Swissmedic).
  SMOFlipid is a white oily emulsion containing soya oil and medium chain triglycerides as main active components, normally used as parenteral nutrition as complement for essential fat acids supplementation. In this study the "white" test (= the administration of SMOFlipid retrograde through the cystic duct) is made by injection of one or two 20cc syringes full of lipidic solution (SMOFlipid 20%) in the cystic stump, directing the flow to the intrahepatic ducts. Residual fat emulsion is washed out from the biliary tract by a low pressure infusion of 20 to 50 ml of saline solution.
  Interventions: Drug: "white" test" (= the administration of SMOFlipid retrograde through the cystic duct)
- Control Intervention (No Intervention): Open bile ducts are identified in the control group by visual control of the liver resection surface combined with the use of white gauzes (standard procedure)

INTERVENTIONS:
Drug: "white" test" (= the administration of SMOFlipid retrograde through the cystic duct) — "white" test" (= the administration of SMOFlipid retrograde through the cystic duct)
  Arms: Experimental Intervention (treatment)

SUMMARY:
Bile leakage (BL) is the most frequent complication after liver resection. This study is to investigate the role of intraoperative administration of SMOFlipid 20% (fat emulsion which allows intraoperative identification of open bile ducts at the liver resection surface when it is administered retrograde through the cystic duct) in terms of prevention of postoperative BL within 30 days after surgery.

DETAILED DESCRIPTION:
Bile leakage (BL) is the most frequent complication after liver resection leading to the need of interventional drainage, endoscopic retrograde cholangio pancreatography (ERCP) or even reoperation. Strategies leading to a reduction of the rate of this complication are valuable. SMOFlipid 20% is a fat emulsion which is primary indicated for parenteral nutrition. Because of its fatty content this solution is white. This allows the clear intraoperative identification of open bile ducts at the liver resection surface when it is administered retrograde through the cystic duct. Consequently, open bile ducts can be sutured preventing the postoperative development of BL. If the rate of bile leakages can be reduced, resources for interventions and relaparotomy will be saved. This study is to investigate intraoperative administration of SMOFlipid 20% in terms of prevention of BL within 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive an anatomical resection of two or more liver segments for any reason with simultaneous cholecystectomy in elective Setting
* Patients who will receive an anatomical resection of two or more liver segments for any reason which already had a cholecystectomy if intraoperatively the cystic stump can be identified and opened
* Ability of subject to understand character and individual consequences of the clinical Trial
* Informed consent documented by signature

Exclusion Criteria:

* Previous cholecystectomy if intraoperative it is not possible to identify the cystic stump
* Intraoperative hepatico-jejunostomy
* Hypersensitivity to fish-, egg-, soybean or peanut protein or to any of the active ingredients or excipients
* Immunosuppression, pregnancy
* Emergency liver resection because of traumatic liver rupture
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
rate of postoperative bile leakage | within 30 days postoperative
  Comparison of the rate of postoperative bile leakage in the control and in the intervention group. This is a binary endpoint defined by the presence or absence of the bile leakage (yes or no). Bile leakage is defined as bilirubin concentration in the drain fluid at least 3 times the serum bilirubin concentration on or after postoperative day 3.

SECONDARY OUTCOMES:
Severity of the bile leakage (Grade A, B or C according to the definition by Koch et al). | within 30 days postoperative
  The severity of bile leakage is classified according to its impact on patients´ clinical management. Grade A bile leakage causes no change in patients' clinical management. A Grade B bile leakage requires active therapeutic intervention but is manageable without relaparotomy, whereas in Grade C bile leakage relaparotomy is required.
In-hospital mortality other than related to the bile leakage | within 30 days postoperative
  In-hospital mortality other than related to the bile leakage
In-Hospital morbidity other than related to the bile leakage | within 30 days postoperative
  In-Hospital morbidity other than related to the bile leakage
Endoscopic retrograde cholangio pancreatography (ERCP) (yes/no) | within 30 days postoperative
  Endoscopic retrograde cholangio pancreatography (ERCP) (yes/no)
Percutaneous Transhepatic Cholangio Drainage (PTCD) (yes/no) | within 30 days postoperative
  Percutaneous Transhepatic Cholangio Drainage (PTCD) (yes/no)
Interventional drainage (yes/no) | within 30 days postoperative
  Interventional drainage (yes/no)
Re-operation (yes/no) | within 30 days postoperative
  Re-operation (yes/no)
Intensive care unit (ICU) stay (in days) | within 30 days postoperative
  Intensive care unit (ICU) stay (in days)
Total hospital stay (in days) | within 30 days postoperative
  Total hospital stay (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Manzini, Dr. med., Principal Investigator — Cantonal Hospital of Aarau, Switzerland
Locations (5):
- Switzerland (5):
  - Department of Visceral Surgery, Cantonal Hospital of Aarau, Aarau
  - Clarunis Basel, Universitäres Bauchzentrum Basel, Basel
  - Kantonsspital Luzern, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen

REFERENCES:
- [Derived] Cristaudi A, Tarantino I, Scheiwiller A, Wiencierz A, Majno-Hurst P, Schmied BM, Metzger J, Hartel M, Kremer M, Manzini G. Diagnostic role of the 'white test' with lipidic solution in the early intraoperative identification of open bile ducts for the prevention of bile leakage after liver resection: study protocol for a randomised controlled multicentric superiority trial (BiLe-Trial). BMJ Open. 2021 Jul 29;11(7):e049449. doi: 10.1136/bmjopen-2021-049449. PMID 34326053